CLINICAL TRIAL: NCT02703363
Title: Minocycline and Celecoxib as Adjunctive Treatments of Bipolar Depression: A Factorial Design Randomised Controlled Trial
Brief Title: Minocycline and Celecoxib as Adjunctive Treatments of Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: Dow University of Health Sciences (Other); Abbasi Shaheed Hospital (Other); Rawalpindi Medical College, Pakistan (Other); University of Manchester (Other); Stanley Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIN-BPD
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Depression; Bipolar Disorder; Bipolar Depression; Mood Disorders
MeSH Terms: conditions — Depression; Bipolar Disorder; Mood Disorders | interventions — Minocycline; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- Minocycline with TAU (Experimental)
  Interventions: Drug: Minocycline
- Celecoxib with TAU (Experimental)
  Interventions: Drug: Celecoxib
- Minocycline and celecoxib with TAU (Experimental)
  Interventions: Drug: Minocycline; Drug: Celecoxib
- Placebo with TAU (Active Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Minocycline
  Arms: Minocycline and celecoxib with TAU; Minocycline with TAU
Drug: Celecoxib
  Arms: Celecoxib with TAU; Minocycline and celecoxib with TAU
Drug: Placebo
  Arms: Placebo with TAU

SUMMARY:
Bipolar disorder is a leading cause of disability worldwide. A high proportion of patients with bipolar disorder experience persistent depressive symptoms that do not respond to standard drug treatments. Recent evidence has suggested that anti-inflammatory treatment may reduce depressive symptoms. Minocycline is a tetracycline antibiotic with good central nervous system (CNS) penetration that has been suggested to be effective as an adjunct drug in improving depressive symptoms. Celecoxib, a selective cyclooxygenase 2 (COX-2) inhibitor, has also shown promising results in the treatment of depressive symptoms. In this factorial design, double blind, randomised controlled trial the investigators will determine the efficacy of minocycline and/or celecoxib as an adjunct to treatment as usual (TAU) in patients experiencing a depressive phase of bipolar I or II disorder. The investigators hypothesise that augmentation with minocycline and/or celecoxib will lead to an improvement in depressive symptoms in participants in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years;
* Diagnostic and Statistical Manual-5 (DSM 5) diagnosis of bipolar I or II disorder and current major depressive disorder;
* Experiencing current depressive symptoms for at least 4 weeks (HAMD-17 score ≥18);
* Competent and willing to give informed consent;
* Taking the current medication for a minimum of 4 week prior to baseline;
* Able to take oral medication;
* If female, willing to use adequate contraceptive precautions and to have monthly pregnancy tests.

Exclusion Criteria:

* Relevant medical illness (HIV, renal, hepatic, cardiac, serious dermatological disorders such as exfoliative dermatitis, systemic lupus erythematosis);
* Prior history of intolerance to any of the tetracyclines or NSAIDs;
* Concomitant penicillin therapy;
* Concomitant anticoagulant therapy;
* Presence of a seizure disorder;
* Currently taking other antibiotics, other NSAIDs, acetazolamide, or methotrexate;
* Any change of psychotropic medications within the previous 4 weeks;
* Diagnosis of substance abuse (except nicotine or caffeine) or dependence within the last 3 months according to DSM-5 criteria;
* Pregnant or breast-feeding;
* Presence of primary psychotic disorder;
* Serious risk of suicide;
* Current three or more manic/hypomanic symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale scores | 12 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- Pakistan (4):
  - Dow University of Health Sciences, Karachi, Sindh
  - Institute of Behavioural Sciences, Karachi, Sindh
  - Karwan-e-Hayat, Karachi, Sindh
  - Abbasi Shaheed Hospital, Karachi, Sindh

REFERENCES:
- [Derived] Husain MI, Chaudhry IB, Khoso AB, Husain MO, Hodsoll J, Ansari MA, Naqvi HA, Minhas FA, Carvalho AF, Meyer JH, Deakin B, Mulsant BH, Husain N, Young AH. Minocycline and celecoxib as adjunctive treatments for bipolar depression: a multicentre, factorial design randomised controlled trial. Lancet Psychiatry. 2020 Jun;7(6):515-527. doi: 10.1016/S2215-0366(20)30138-3. Epub 2020 May 20. PMID 32445690